CLINICAL TRIAL: NCT01516684
Title: A Randomized, Double Blind Trial of Pediatric Lumbar Puncture Under Sedation/Total Intravenous Anesthesia (TIVA) With and Without EMLA Cream
Brief Title: Local Anesthetic Cream in Younger Patients Undergoing Lumbar Punctures
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IRB00017079; NCI-2012-00019 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCCWFU 01211 (Other: Wake Forest University Health Sciences)
Record Dates: First submitted 2012-01-20; First posted 2012-01-25 (Estimated); Results first posted 2019-09-06 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-08

CONDITIONS: Malignant Neoplasm
MeSH Terms: conditions — Neoplasms | interventions — Lidocaine, Prilocaine Drug Combination; Propofol; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (EMLA) (Experimental): Patients receive topical EMLA cream 60 minutes to 4 hours prior to the LP followed by standard sedation with fentanyl citrate and propofol.
  Interventions: Drug: EMLA; Drug: propofol; Drug: fentanyl citrate
- Arm II (placebo) (Active Comparator): Patients receive topical placebo cream 60 minutes to 4 hours prior to the LP followed by standard sedation with fentanyl citrate and propofol.
  Interventions: Drug: placebo administration; Drug: propofol; Drug: fentanyl citrate

INTERVENTIONS:
Drug: placebo administration — Given topically
  Arms: Arm II (placebo)
Drug: EMLA — Given topically
  Other Names: eutectic mixture of local anesthetics; lidocaine-prilocaine; lidocaine-prilocaine eutectic mixture
  Arms: Arm I (EMLA)
Drug: propofol — Given IV
  Other Names: Diprivan
Drug: fentanyl citrate — Given IV
  Other Names: Actiq; Oralet; Sublimaze

SUMMARY:
This randomized clinical trial studies local anesthetic (EMLA) cream in younger patients undergoing lumbar punctures (LP). A local anesthetic cream may be effective for numbing the skin and reducing movement when applied prior to lumbar punctures and may reduce the amount of sedation necessary

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether the application of a topical anesthetic (EMLA cream) to the LP site will decrease the total dose of propofol administered to pediatric oncology patients who are being sedated for LPs compared to application of a topical placebo cream.

SECONDARY OBJECTIVES:

I. To determine whether the use of EMLA cream decreases complication rates from sedation.

II. To determine whether the use of EMLA cream decreases traumatic lumbar punctures.

III. To determine whether the use of EMLA cream shortens recovery time. IV. To determine practitioner and parent satisfaction with the use of EMLA cream.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive topical EMLA cream 60 minutes to 4 hours prior to the LP followed by standard sedation with fentanyl citrate and propofol.

ARM II: Patients receive topical placebo cream 60 minutes to 4 hours prior to the LP followed by standard sedation with fentanyl citrate and propofol.

After completion of study treatment, patients are followed up within 1 week.

ELIGIBILITY:
Inclusion Criteria:

Pediatric oncology patients undergoing a lumbar puncture in the Pediatric Sedation Suite; patients may or may not be receiving intrathecal chemotherapy

Exclusion Criteria:

Patients undergoing additional procedures during the same anesthetic such as bone marrow aspirate or biopsy will be excluded because they will likely require higher doses of propofol than those undergoing LP alone Patients who are allergic to or not tolerant of EMLA cream, propofol, or fentanyl will be excluded Patients who are pregnant will be excluded Patients having their LPs done by students will be excluded

Max Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 33 (Actual)
Dates: Start 2012-05-14 (Actual); Primary Completion 2018-06-26 (Actual); Study Completion 2018-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dudley Hammon, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Originally 33 participants were registered, with 170 trials; each participant had between 1-14 trials (median=4).
  Five of these participants did not end up receiving the procedure and 1 was a screen fail, leaving 27 participants with between 1-14 trials (median=5).
Units Other Than Participants: Trials
Groups:
- Arm A (EMLA): Patients receive topical EMLA cream 60 minutes to 4 hours prior to the lumbar puncture followed by standard sedation
- Arm B (Placebo): Patients receive topical placebo cream 60 minutes to 4 hours prior to the LP followed by standard sedation
Period: Overall Study
Arm/Group | Arm A (EMLA) | Arm B (Placebo)
Started | NA; 85 Trials (Overall number of units (trials) was used for measuring results with 170 trials. Trials were randomized for each arm, not participants) | NA; 85 Trials (Overall number of units (trials) was used for measuring results with 170 trials. Trials were randomized for each arm, not participants)
Completed (Overall number of units (trials) completed was 152) | NA; 75 Trials (Trials were randomized for each arm, not participants) | NA; 77 Trials (Overall number of units (trials) completed was 152 Trials were randomized for each arm, not participants)
Not Completed | NA; 10 Trials | NA; 8 Trials

BASELINE CHARACTERISTICS:
Population: Participants were not randomized to the arms. The trials for each arm were randomized so we are using the trials to report demographics by arm.
Units Other Than Participants: Trials
Groups:
- Arm A (EMLA): Trials completed is the unit of measure, not participants.
  Patients receive topical EMLA cream 60 minutes to 4 hours prior to the lumbar puncture followed by standard sedation
- Arm B (Placebo): Trials completed is the unit of measure, not participants.
  Patients receive topical placebo cream 60 minutes to 4 hours prior to the LP followed by standard sedation
- Total: Total of all reporting groups
Arm/Group | Arm A (EMLA) | Arm B (Placebo) | Total
Number analyzed (Participants) | NA | NA | NA
Number analyzed (Trials) | 75 | 77 | 152
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.7 (5.4) | 8.8 (5.3) | 8.2 (5.4)
Sex: Female, Male [Count of Units; unit: Trials]
  Female | 22 | 22 | 44
  Male | 53 | 55 | 108
Ethnicity (NIH/OMB) [Count of Units; unit: Trials] — Participants were not randomized, the trials were randomized so we are using the trials (completed) to report demographics by arm
  Trials
    Hispanic or Latino | 10 | 10 | 20
    Not Hispanic or Latino | 65 | 67 | 132
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Units; unit: Trials] — Participants were not randomized, the trials were randomized so we are using the trials (completed) to report demographics by arm
  Trials
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 14 | 18 | 32
    White | 60 | 56 | 116
    More than one race | 1 | 3 | 4
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: Trials completed] — Participants were not randomized, the trials were randomized so we are using the trials (completed) to report demographics by arm
  Trials completed
    United States | 75 | 77 | 152

OUTCOME MEASURES:

1. Primary Outcome: Total Dose of Propofol Administered to Each Patient
Description: Analyzed using descriptive statistics and mixed model regression methods. Raw mean total dose administered and raw percentage of times additional propofol was administered will be presented by sedation group treating each event (sedation with lumbar puncture) as the unit. T-test and chi-square tests will be performed as appropriate.
Time Frame: 20 minutes after sedation
Population: Participants were not randomized. Trials were randomized so we will have to use the trials to report by arm
Measure: Least Squares Mean (Standard Error); unit: mg/kg
Units Other Than Participants: Trials
Arm/Group | Arm A (EMLA) | Arm B (Placebo)
Number analyzed (Participants) | NA | NA
Number analyzed (Trials) | 75 | 77
mg/kg | 2.94 (0.25) | 3.22 (0.19)
Statistical Analysis 1: Comparison: Arm A (EMLA) vs Arm B (Placebo); Raw mean total dose administered and raw percentage of times additional propofol was administered will be presented by sedation group treating each event (sedation with lumbar puncture) as the unit. T-test and chi-square tests will be performed as appropriate for the outcome. GEE methods will be used when analyzing the percentage of times additional propofol was administered. Mixed model regression methods will be used when analyzing the total dose administered; Test type: Other; p = 0.036, T-test and chi-square

2. Secondary Outcome: Level of Movement (no Movement, Minor Movement, Major Movement, Other) After EMLA Cream or Placebo Cream Administration
Time Frame: At the time of LP insertion
Population: Participants were not randomized. Trials were randomized so we will use the trials to report by arm
Measure: Count of Units; unit: Trials
Units Other Than Participants: Trials
Arm/Group | Arm A (EMLA) | Arm B (Placebo)
Number analyzed (Participants) | NA | NA
Number analyzed (Trials) | 75 | 77
Trials
  No movement | 50 | 29
  Minor movement | 7 | 12
  Major movement | 8 | 27
  Other | 10 | 9

3. Secondary Outcome: Complications Including Any Change in Vital Signs That Requires Intervention by the Sedation Team, as Well as Post-LP Headache From Sedation With or Without EMLA Cream
Description: Each patient's parent (and/or the patient) will be contacted by telephone within one week of the lumbar puncture (or in person if the next clinic visit is within one week) to ask if the patient had any headache after the lumbar puncture, and if they had any other complications.
Time Frame: Within one week of the LP
Population: Not all procedures were completed at all trials. Participants were not randomized. Trials were randomized so will use the trials to report by arm.
Measure: Mean (Standard Error); unit: Probability of experiencing headache
Units Other Than Participants: Trials
Arm/Group | Arm A (EMLA) | Arm B (Placebo)
Number analyzed (Participants) | NA | NA
Number analyzed (Trials) | 68 | 73
Probability of experiencing headache | 0.194 (0.041) | 0.289 (0.057)
Statistical Analysis 1: Comparison: Arm A (EMLA) vs Arm B (Placebo); Test type: Other — Marginal mixed model (GEE type); p = 0.094, Mixed Models Analysis

4. Secondary Outcome: Traumatic Lumbar Punctures After EMLA Cream or Placebo Cream Administration
Description: Traumatic lumbar puncture is defined as lumbar puncture in which cerebrospinal fluid contains at least 10 red blood cells (RBCs) per microliter and bloody lumbar as one in which the cerebrospinal fluid contained at least 500 red blood cells (RBCs) per microliter.
Time Frame: 20 minutes after lumbar puncture
Population: Total number of trials was 136, 15 are missing. Participants were not randomized. Trials were randomized so will use the trials to report by arm.
Measure: Count of Units; unit: Trials
Units Other Than Participants: Trials
Arm/Group | Arm A (EMLA) | Arm B (Placebo)
Number analyzed (Participants) | NA | NA
Number analyzed (Trials) | 70 | 66
Trials
  Atraumatic | 63 | 57
  Traumatic | 6 | 5
  Bloody | 1 | 4
Statistical Analysis 1: Comparison: Arm A (EMLA) vs Arm B (Placebo); Test type: Other; p = 0.382, Chi-squared

5. Secondary Outcome: Complications Including Any Change in Vital Signs That Requires Intervention by the Sedation Team, Post-LP Back Pain From Sedation With or Without EMLA Cream
Description: Each patient's parent (and/or the patient) will be contacted by telephone within one week of the lumbar puncture (or in person if the next clinic visit is within one week) to ask if the patient had any back pain after the lumbar puncture, and if they had any other complications.
Time Frame: Within one week of the LP
Population: as for outcome 3
Measure: Mean (Standard Error); unit: Probability of experiencing back pain
Units Other Than Participants: Trials
Arm/Group | Arm A (EMLA) | Arm B (Placebo)
Number analyzed (Participants) | NA | NA
Number analyzed (Trials) | 69 | 74
Probability of experiencing back pain | 0.211 (0.049) | 0.250 (0.054)
Statistical Analysis 1: Comparison: Arm A (EMLA) vs Arm B (Placebo); Test type: Other — Marginal mixed model (GEE type); p = 0.426, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: Up to one week after lumbar puncture
Description: The principal investigator reports there were no adverse events during the randomized trials.
Arm/Group | Arm A (EMLA) | Arm B (Placebo)
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/77
Serious Adverse Events (participants affected / at risk) | 0/75 | 0/77
Other Adverse Events (participants affected / at risk) | 0/75 | 0/77

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2015-08-26): https://cdn.clinicaltrials.gov/large-docs/84/NCT01516684/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2012-07-19): https://cdn.clinicaltrials.gov/large-docs/84/NCT01516684/Prot_SAP_001.pdf